CLINICAL TRIAL: NCT05016518
Title: Comparison of Quality of Recovery (QoR)-15 Scores According to the Use of Anesthetics During Total Intravenous Anesthesia in Female Patients Undergoing Thyroid Surgery
Brief Title: Comparison of Quality of Recovery (QoR)-15 Scores Between Propofol and Remimazolam Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Young Song, Associate professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-0424-002
Record Dates: First submitted 2021-08-10; First posted 2021-08-23 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Patients Undergoing Thyroid Surgery for Neoplasm

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol group (Experimental): Propofol based total intravenous anesthesia
  Interventions: Drug: Arm I (Propofol group)
- Remimazolam group (Active Comparator): Remimazolam based total intravenous anesthesia
  Interventions: Drug: Arm II (Remimazolam group)

INTERVENTIONS:
Drug: Arm I (Propofol group) — Propfol group will be started and maintained total intravenous anesthesia with propofol and remifentanil .
  Arms: Propofol group
Drug: Arm II (Remimazolam group) — Remimazolam group will be started and maintained total intravenous anesthesia with remimazolam and remifentanil.
  Arms: Remimazolam group

SUMMARY:
Remimazolam is a ultra-short-acting benzodiazepine that is rapidly metabolized in the body by tissue esterase and not accumulates in the body for long periods of infusion. In addition, similar to other benzodiazepines, it is possible to reverse the sedation and anesthetic effects through flumazenil. It has no injection pain and infusion syndrome compared with propofol. There is no study to investigate overall postoperative functional recovery via QoR-15 in patients receiving TIVA using remimazolam. The purpose of this study is to determine whether there is any difference in the quality of postoperative recovery between propofol-based and remimazolam-based total intravenous anesthesia in female patients undergoing thyroidectomy. The QoR-15 questionnaire score, pain, nausea/vomiting, and the frequency of complications are evaluated and compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

•20≤Age≤65 female Open thyroidectomy ASA-PS I-III

Exclusion Criteria:

* Allergic history of any study drug
* Taking any sedative, opioid, or sleep aid drugs
* Psychiatric or neurological disorder
* BMI>30 kg/m2
* Pregnancy
* Vulnerable patients

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
postoperative day 1(POD1) Quality of Recovery(QoR)-15 questionnaire score | Postoperative day 1
  Quality of life will be evaluated using Quality of Recovery(QoR)-15 questionnaire score at postoperative day 1(minimum value : 0, maximum value : 150, the higher the score, the better the result)

SECONDARY OUTCOMES:
postoperative day 2(POD2) Quality of Recovery(QoR)-15 questionnaire score | Postoperative day 2
  Quality of life will be evaluated using Quality of Recovery(QoR)-15 questionnaire score at postoperative day 2(minimum value : 0, maximum value : 150, the higher the score, the better the result)
Response time | perioperative - until 48hours
  Time from cessation of main anaesthetics to patients' response to verbal command
Tracheal extubation time | perioperative - until 48hours
  Time from cessation of main anaesthetics to tracheal extubation
Time to recovery of self respiration | perioperative - until 48hours
  Time from cessation of main anaesthetics to recovery of spontaneous breathing
PACU(post-anesthesia care unit) stay time | perioperative - until 48hours
  from entry of PACU to go general ward
Postoperative pain score | at admission to PACU, discharge from PACU, postoperative 6hours
  postoperative pain score measured by 11-point NRS(numerical rating scale) score (minimum : 0, maximum : 11, the lower the score, the lesser pain)
Postoperative nausea and vomiting | at admission to PACU, discharge from PACU, postoperative 6hours
  postoperative nausea and vomiting will be evaluated using 2 point scale (yes, no) at admission to PACU, discharge from PACU, postoperative 6hours
Postoperative sedation score | at admission to PACU, discharge from PACU
  monitored through the sedation scale called Richmond Agitation-Sedation Scale(RASS). RASS is a medical scale used to measure the agitation or sedation level of a person.The score ranges from +4 "combative" to -5 "unarousable".
the incidence of administration of postoperative rescue drug | perioperative - until 72hours
  administration of analgesic drug and anti-emetic drug for postoperative management
hospital stay | preoperative - until discharge (usually 48 hours to 72hours)
  days of hospital stay
postoperative complications | preoperative - until discharge (usually 48 hours to 72hours)
  postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Young Song, Principal Investigator — GangnamSeverance Hospital
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea